CLINICAL TRIAL: NCT05918016
Title: Ultrasonographic Prognostic Scale of Periventricular Hemorrhagic Infarction in Preterm Infants With Gestational Age <30 Weeks
Brief Title: Ultrasonographic Prognostic Scale of Periventricular Hemorrhagic Infarction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Manuel Sanchez Luna (Other)
Responsible Party: Sponsor-Investigator, Manuel Sanchez Luna, Doctor, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Other Study IDs: Neuro.Neo.1.IVH
Record Dates: First submitted 2023-06-07; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Preterms; Infarction Cerebral
MeSH Terms: conditions — Cerebral Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Routine cranial ultrasounds — we will use the routine cranial ultrasounds

SUMMARY:
Observational study of preterm infant with a gestational age < 30 weeks born between 2017-2023 in Neonatal Care Unit in Gregorio Marañon Hospital (Madrid, Spain). We use a new ultrasonographic prognostic scale of periventricular hemorrhagic infarction for neurodevelopmental outcome at age 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Gestacional Age < 30 weeks

Exclusion Criteria:

* Brain malformation
* Genetic syndrome
* Metabolic disorders
* Chromosomal abnormality
* None cranial ultrasound

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newborn with gestational age < 30 weeks
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Periventricular Hemorrhagic Infarction | first month
  Yes or no
Characteristic Sonographic | first month
Neurodevelopmental outcome at age 2 years | first month

SECONDARY OUTCOMES:
Medical records | first month

CONTACTS AND LOCATIONS:
Locations (1):
- Gregorio Marañon Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No